CLINICAL TRIAL: NCT07399197
Title: Three-Dimensional Evaluation of Alveolar Bone Changes and Root Resorption After Orthodontic Traction of Unilateral Buccally Displaced Maxillary Canines Using Two Different Techniques: A Randomized Clinical Trial
Brief Title: 3-D Evaluation of Alveolar Bone Changes and Root Resorption BDMC
Acronym: BDMC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Mohammed Abdullah Abdullah Al-Hababy, Candidate in PhD of Orthodontics, Sana'a University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR:04/03/2025
Record Dates: First submitted 2026-01-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion; Displaced Teeth
Keywords: Buccally Displaced Maxillary Canines; Alveolar Bone Changes; Root Resorption; Orthodontic Treatment
MeSH Terms: conditions — Malocclusion; Root Resorption

STUDY DESIGN:
Intervention Model Description: This clinical trial will use a randomized design with equal allocation in a 1:1 ratio, blinding, and paralleling two groups. The study will compare the treatment outcomes between the segmental T-loop and the piggyback double wire traction techniques.
  The study will use CBCT images to evaluate the 3-D changes in the alveolar bone and root length of the unilateral BDMCs and adjacent teeth before and after orthodontic traction and compare them with the normal contralateral canines and adjacent teeth.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: This clinical trial will use a randomized design with equal allocation in a 1:1 ratio, blinding, and paralleling two groups.Computer-generated random sequencing using Microsoft Office Excel will performed. Opaque sealed envelopes will be used for allocation concealment. Blinding of the participants and operator will not possible because of the nature of the study. Blinding of the result evaluation will be done through data concealment during assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-loop (Active Comparator): In patients randomized to the frictionless group, T-loops were fabricated using 0.017 X 0.025-inch TMA wire.
  The posterior leg of the T-loops will be inserted in the auxiliary tube of the first molar, and the anterior leg engaged the canine bracket.
  Interventions: Device: T-loop
- Piggyback double wire (Active Comparator): In patients randomized to the piggyback double wire method, all teeth in both maxillary and mandibular arches will be bonded with preadjusted edgewise brackets from the 0.022- in-slot MBT system.
  Interventions: Device: Piggyback double wire

INTERVENTIONS:
Device: T-loop — Firstly, only the BDMC will be bonded with a preadjusted edgewise bracket from the 0.022-in-slot MBT system and cementing the trans palatal arch.
  Canine traction will be carried out by ligating the segmental T loop of 0.016×0.022 TMA wire on the BDMC and inserting the other end of the T loop in the maxillary first permanent molar tube. The segmented T loop will be activated by 2 mm per month and tightened posteriorly to the tube of the first permanent molar for approximately 3 months to move the canine.
  Once the BDMC is in the proper site in the maxillary arch, all teeth in both maxillary and mandibular arches will be bonded with preadjusted edgewise brackets from the 0.022-in-slot MBT system. Leveling and alignment will start with engaging 0.014-in NiTi arch wires in both arches.
  Arms: T-loop
Device: Piggyback double wire — All teeth in both maxillary and mandibular arches will be bonded with preadjusted edgewise brackets from the 0.022- in-slot MBT system. Leveling and alignment will start with engaging 0.014-in NiTi arch wires in both arches, bypassing maxillary BDMC.
  The arch wire sequence will include 0.014-in NiTi, 0.016-inch NiTi, 0.016x0.022-inch NiTi.
  After the arches are properly aligned, the piggyback technique will be used on the maxillary arch, and the arch wire size will be increased to 0.016 x 0.016-inch stainless15 steel for the maxillary arch and ligating the accessory 0.012-inch NiTi round for BDMC traction.
  Arms: Piggyback double wire

SUMMARY:
This clinical study used CBCT images to investigate the alveolar bone changes and root resorption in unilateral buccally displaced maxillary canines and adjacent teeth before and after orthodontic traction of unilateral BDMCs.

The CBCT images will also be used to compare these changes to the normal contralateral side. The study outcome is to compare the 3-D changes in the alveolar bone and dental roots between the 2 interventional techniques (segmentalT-loop and piggyback NiTi traction) methods.

DETAILED DESCRIPTION:
Buccally displaced eruptions of permanent maxillary canines occur in 0.8% to 5.2% of orthodontic cases. Patients are often motivated to request orthodontic treatment when they have crowded teeth and maxillary canines that come in buccally erupted.

The treatment of BDMC is challenging due to the limited labial alveolar bone and the potential risks of root resorption, bone loss, and gingival recession due to the movement of long and bulge roots, necessitating bodily movement with light and constant orthodontic force. The previous studies focused only on comparisons of root resorption, bone loss, and periodontal health before and after impacted canine traction. The previous studies on BDMC mainly included case reports that looked at various orthodontic traction methods. To our knowledge, no randomized clinical trial has been done to study the 3- D changes in the alveolar bone and root length after orthodontic traction of BDMCs.

ELIGIBILITY:
Inclusion Criteria:

* Yemeni ethnic patients.
* Presence of unilateral BDMC.
* The presence of a properly positioned and normally erupted contralateral canine.
* Mild to moderate crowding.
* The need for fixed orthodontic treatment.
* No sagittal discrepancy

Exclusion Criteria:

* History of severe facial trauma.
* Previous orthodontic treatment.
* Presence of bilateral BDMC.
* Presence of developmental dental anomalies.
* Presence of facial syndromes and bone metabolism disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in the Alveolar Bone Thickness | From baseline (before orthodontic traction) to the completion of orthodontic traction (an average of 8 months)
  The mean change in the alveolar bone thickness will be measured in millimeters (mm) using CBCT scans.
Mean Change in the Alveolar Bone Height | Baseline and Month 8
  Alveolar bone height measured in millimeters (mm) using CBCT.

SECONDARY OUTCOMES:
Mean Change in Root Resorption | Baseline and Month 8
  The rate of external root resorption in mm measured using CBCT scans.
Difference Between Two groups in Alveolar Bone Dimension Changes | Month 8 after the completion of canine traction.
  Measuring the mean change in alveolar bone dimension (mm) between Segmental T loop and Piggyback Orthodontic traction techniques using CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Al-Hababy, MSC, Principal Investigator — Sana'a University

IPD SHARING:
Plan to Share IPD: No